CLINICAL TRIAL: NCT02342756
Title: Esophageal Pressure-Guided Optimal PEEP/mPaw in CMV and HFOV: The EPOCH Study
Acronym: EPOCH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Toronto (Other)
Collaborators: University Health Network, Toronto (Other); Nihon Kohden (Industry)
Responsible Party: Principal Investigator, Eddy Fan, Eddy Fan, MD, PhD, Assistant Professor of Medicine, Interdepartmental Division of Critical Care Medicine, University of Toronto
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 14-8253
Record Dates: First submitted 2015-01-15; First posted 2015-01-21 (Estimated); Last update posted 2015-01-30 (Estimated); Status verified 2015-01

CONDITIONS: Respiratory Distress Syndrome, Adult; Ventilator-Induced Lung Injury
Keywords: ARDS, HFOV
MeSH Terms: conditions — Respiratory Distress Syndrome; Ventilator-Induced Lung Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1: CMV - HFOV (Experimental): Patients in group 1 will start with conventional mechanical ventilation with different values of PEEP (A-PEEP so that PLEEO = 0 cmH2O, B- PEEP so that PLEIO = 15 cmH2O, C- PEEP so that PLEEO = 0 cmH2O) and then will be ventilated with high frequency oscillatory ventilation (D- mPaw so that PL = 0 cmH2O, E- mPaw so that PL = 15 cmH2O, F- mPaw so that PL = 0 cmH2O)
  Intervention: Device: Targeting transpulmonary pressure to avoid VILI
  Interventions: Device: Targeting transpulmonary pressure to avoid VILI
- Group 2: HFOV - CMV (Experimental): Patients in group 2 will start with high frequency oscillatory ventilation (D- mPaw so that PL = 0 cmH2O, E- mPaw so that PL = 15 cmH2O, F- mPaw so that PL = 0 cmH2O) and then will be ventilated with conventional mechanical ventilation with different values of PEEP (A-PEEP so that PLEEO = 0 cmH2O, B- PEEP so that PLEIO = 15 cmH2O, C- PEEP so that PLEEO = 0 cmH2O).
  Intervention: Device: Targeting transpulmonary pressure to avoid VILI
  Interventions: Device: Targeting transpulmonary pressure to avoid VILI

INTERVENTIONS:
Device: Targeting transpulmonary pressure to avoid VILI — Set different values of PEEP (CMV) and mPaw (HFOV) to obtain determined values of transpulmonary pressure (0 and 15 centimeters of water) and to determine the impact of ventilation on VILI

SUMMARY:
The use of positive end-expiratory pressure (PEEP) has been shown to prevent the cycling end-expiratory collapse during mechanical ventilation and to maintain alveolar recruitment, keeping lung portions open, increasing the resting end-expiratory volume. On the other hand PEEP may also overdistend the already open lung, increasing stress and strain.

Theoretically high frequency oscillatory ventilation (HFOV) could be considered an ideal strategy in patients with ARDS for the small tidal volumes, but the expected benefits have not been shown yet.

PEEP and HFOV should be tailored on individual physiology. Assuming that the esophageal pressure is a good estimation of pleural pressure, transpulmonary pressure can be estimated by the difference between airway pressure and esophageal pressure (PL= Paw - Pes). A PL of 0 cmH2O at end-expiration should keep the airways open (even if distal zones are not certainly recruited) and a PL of 15 cmH2O should produce an overall increase of lung recruitment.

The investigators want to determine whether the prevention of atelectrauma by setting PEEP and mPaw to obtain 0 cmH2O of transpulmonary pressure at end expiratory volume is less injurious than lung recruitment limiting tidal overdistension by setting PEEP and mPaw at a threshold of 15 cmH2O of transpulmonary pressure.

The comparison between conventional ventilation with tidal volume of 6 ml/Kg and HFOV enables us to understand the role of different tidal volumes on preventing atelectrauma and inducing lung recruitment.

The use of non-invasive bedside techniques such as lung ultrasound, electrical impedance tomography, and transthoracic echocardiography are becoming necessary in ICU and may allow us to distinguish between lung recruitment and tidal overdistension at different PEEP/mPaw settings, in order to limit pulmonary and hemodynamic complications during CMV and HFOV.

DETAILED DESCRIPTION:
The absolute value of esophageal pressure (Pes), measured during an end-expiratory pause can be considered a good surrogate for pleural pressure (Ppl), and the difference between airway pressure (Paw) and Pes a valid estimation of transpulmonary pressure (PL). Although this method has not been tested in large clinical trials yet, the utility of Pes in guiding therapy of ARDS has been shown in EPVent study.

Therefore, assuming that Pes is a good estimation of Ppl, PEEP and mPaw could be targeted to obtain different value of PL. A PL of 0 cmH2O at end-expiratory pause, should keep the airways open (even if distal zones are not certainly recruited) and a PL of 15 cmH2O at end-inspiratory pause should produce an overall increase of lung recruitment, limiting tidal overdistension. The comparison of these two different ventilatory settings allows us to determine whether the prevention of atelectrauma by setting PEEP and Paw of HFOV to obtain 0 cmH2O of transpulmonary pressure at end-expiratory occlusion is less injurious than lung recruitment limiting tidal overdistension by setting PEEP and mPaw at a threshold of 15 cmH2O of transpulmonary pressure.

The use of HFOV beside conventional ventilation, enables us to understand the role of these ventilatory strategies with different end-expiratory volumes, on preventing atelectrauma and inducing lung recruitment.

In addition the use of non-invasive bedside techniques as pleural and lung ultrasonography (PLUS), electrical impedance tomography (EIT), and transthoracic echocardiography (TTE) may allow us to distinguish between lung recruitment and tidal overdistension at different PEEP/mPaw settings, in order to limit pulmonary and hemodynamic complications during CMV and HFOV, and may help in the assessment of recruitable lungs.

Primary objective:

To determine whether the prevention of atelectrauma by setting PEEP (CMV) to obtain 0 cmH2O of transpulmonary pressure at end-expiratory occlusion and mPaw (HFOV) to obtain 0 cmH2O of mean transpulmonary pressure is less injurious than lung recruitment limiting tidal overdistension by setting PEEP (CMV) and mPaw (HFOV) at a threshold of 15 cmH2O of transpulmonary pressure. Plasma cytokines will be used to define the ventilator induced lung injury.

Secondary objectives:

1. To assess lung recruitment and tidal overdistension with bedside non-invasive methods such as EIT and PLUS during CMV and HFOV, with PEEP and mPaw set to obtain a PL of 0 and a PL of 15 cmH2O.
2. To assess if the impact of PEEP and HFOV set to obtain PL of 15 cmH2O is more dangerous for right ventricular function than PEEP to obtain PLEEO and PLHFOV of 0 cmH2O. TTE will be used to evaluate the heart function.

Study management:

For this pathophysiological study we will enroll 20 patients with moderate or severe ARDS, within 72 hours of arrival in our ICU.

1. All patients will be supine, with the head of the bed elevated to 30 degrees.
2. All patients will be deeply sedated and ventilated according to clinical practice.
3. Monitoring will be provided at least with:

   * Heart rate (HR) and cardiac rhythm.
   * Mean arterial pressure (MAP) monitored by invasive blood pressure via an arterial catheter.
   * Central venous pressure (CVP).
   * Transcutaneous O2 saturation by pulse oximetry (SpO2),
   * Airflow, airway pressure (Paw), tidal volume (Vt), end-tidal partial pressure of carbon dioxide (PETCO2)
4. Immediately before the initiation of the study, the patients will be subjected to neuromuscular blockade with a cisatracurium intravenous bolus and continuous infusion titrated to achieve 0-2/4 twitches on facial nerve electrical stimulation.
5. A nasogastric catheter with esophageal and gastric balloon will be placed. Esophageal pressure (Pes) will be measured during an end-inspiratory (PesEIO) and an end-expiratory occlusion (PesEEO) of the airway. The variation of esophageal pressure during tidal inflation (ΔPes) will be calculated as the difference between PesEIO and PesEEO. Transpulmonary pressure (PL) will be calculated as the difference between Paw and Pes (PL = Paw - Pes). The intragastric pressure will be measured only during an end-expiratory occlusion of the airway (IGP).

All study data will be transcribed directly on to standardized Case Report Forms (CRF).

Patients will be randomized to start the protocol with the controlled mechanical ventilation strategy or the high frequency oscillatory ventilation. A block-randomization scheme with opaque envelopes and block size of 2 will be used.

Study protocol:

Immediately after enrolment, Pes will be measured during an end-expiratory (PesEEO) and end-inspiratory occlusion (PesEIO). PEEP to reach a PLEEO of 0 cmH2O and PEEP to reach a PLEIO of 15 cmH2O will be calculated.

CMV phase A. PLEEO = 0

1. Patients will be ventilated with CMV using the following parameters (in group 2 before starting PesEEO and PesEIO will be measured):

   1. Vt 6 ml/kg predicted body weight
   2. PEEP so that PLEEO = 0 cmH2O
   3. Respiratory Rate (RR) to reach pH 7.25-7.35
   4. FiO2 to have SpO2 ≥ 90%
2. After 40 minutes at these settings, lung ultrasound will be performed to obtain a lung ultrasound score.
3. After completing PLUS, TTE will be performed
4. After completing TTE, EIT will be positioned and recordings of global and regional time courses of impedance changes and associated EIT images will be obtained
5. Blood sample for cytokines measurement will be collected and the following parameters will be measured:

   * Arterial blood gases
   * Crs
   * Alveolar dead space.

B. PLEIO = 15

1. Patients will be ventilated with the same Vt, RR and FiO2 of phase A. PEEP will be set at the value obtained to reach a PLEIO = 15 cmH2O.
2. Same measurements will be repeated as in phase A (steps 2 to 5).

C. PLEEO = 0

1. Patients will be ventilated with the same Vt, RR and FiO2 of previous phases. PEEP will be set at the same value of phase A (PEEP so that PLEEO = 0 cmH2O).
2. Same measurements will be repeated as in phase A (steps 2 to 5). PesEEO and PesEIO will be measured so that CMV phase is completed.

HFOV phase D. PL = 0

1. Patients will be switched to HFOV. Pes will be measured and mPaw to reach a PLHFOV of 0 and of 15 will be calculated. Patients will be ventilated using the following parameters:

   1. Pressure amplitude 90 cmH2O
   2. mPaw to reach a PL of 0 cmH2O
   3. Respiratory Rate (RR) ≥ 5Hz to reach pH 7.25-7.35
   4. FiO2 to have SpO2 ≥ 90%
2. Same measurements will be performed as in phase A (steps 2 to 4). Blood sample for cytokines measurement will be collected and the following parameters will be measured:

   * Arterial blood gases.

E. PL = 15

1. Patients will be ventilated with the same HFOV setting, except for mPaw, which will be set to reach a PL of 15 cmH2O.
2. Same measurements will be performed as in phase D.

F. PL = 0

1. Patients will be ventilated with the same HFOV setting, except for mPaw, which will be set to reach a PL of 0 cmH2O.
2. Same measurements will be performed as in phase D. Then Pes will be measured and HFOV phase is completed.

ELIGIBILITY:
Inclusion Criteria:

* Moderate or severe ARDS, defined according to the Berlin definition (2);
* Endotracheal intubation or tracheostomy

Exclusion Criteria:

* Severe heart failure/cardiogenic shock;
* Pulmonary arterial hypertension requiring systemic vasodilators;
* Contraindications to esophageal balloon: esophageal pathology (stricture, perforation, high grade of varices), recent history of esophageal or gastric surgery, upper GI tract bleeding, severe coagulopathy and nasal trauma;
* Contraindications to Electrical Impedance Tomography (EIT): a temporary or permanent pacemaker, or implantable cardioverter-defibrillator (ICD);
* Age < 16 years.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Ventilator-induced lung injury (VILI) in patients with ARDS as measured by serum cytokines | 1 hour after initiation of each experimental ventilation strategy
  IL-6, TNF, IL-10, IL-1β, and IL-1ra and other cytokines will be detected in EDTA plasma with commercially available enzyme-linked immunosorbent assays (ELISA)

SECONDARY OUTCOMES:
Assessment of lung recruitment and tidal overdistension | 1 hour after initiation of each experimental ventilation strategy
  Lung ultrasound score (LUS), global and regional impedance (EIT).
Impact of transpulmonary pressure on right ventricular function (RV) | 1 hour after initiation of each experimental ventilation strategy
  Measurements: Transthoracic echocardiography (TTE).

CONTACTS AND LOCATIONS:
Overall Officials: Eddy Fan, MD, PhD, Principal Investigator — University Health Network, Toronto; Francesca Facchin, MD, Principal Investigator — University Health Network, Toronto
Locations (2):
- Canada (2):
  - Intensive Care Unit (ICU) of Mount Sinai Hospital, Toronto, Ontario
  - Medical Surgical ICU - Toronto General Hospital, Toronto, Ontario

REFERENCES:
- [Background] Tremblay L, Valenza F, Ribeiro SP, Li J, Slutsky AS. Injurious ventilatory strategies increase cytokines and c-fos m-RNA expression in an isolated rat lung model. J Clin Invest. 1997 Mar 1;99(5):944-52. doi: 10.1172/JCI119259. PMID 9062352
- [Background] Fan E, Needham DM, Stewart TE. Ventilatory management of acute lung injury and acute respiratory distress syndrome. JAMA. 2005 Dec 14;294(22):2889-96. doi: 10.1001/jama.294.22.2889. PMID 16352797
- [Background] Meade MO, Cook DJ, Guyatt GH, Slutsky AS, Arabi YM, Cooper DJ, Davies AR, Hand LE, Zhou Q, Thabane L, Austin P, Lapinsky S, Baxter A, Russell J, Skrobik Y, Ronco JJ, Stewart TE; Lung Open Ventilation Study Investigators. Ventilation strategy using low tidal volumes, recruitment maneuvers, and high positive end-expiratory pressure for acute lung injury and acute respiratory distress syndrome: a randomized controlled trial. JAMA. 2008 Feb 13;299(6):637-45. doi: 10.1001/jama.299.6.637. PMID 18270352
- [Background] Talmor D, Sarge T, Malhotra A, O'Donnell CR, Ritz R, Lisbon A, Novack V, Loring SH. Mechanical ventilation guided by esophageal pressure in acute lung injury. N Engl J Med. 2008 Nov 13;359(20):2095-104. doi: 10.1056/NEJMoa0708638. Epub 2008 Nov 11. PMID 19001507
- [Background] Akoumianaki E, Maggiore SM, Valenza F, Bellani G, Jubran A, Loring SH, Pelosi P, Talmor D, Grasso S, Chiumello D, Guerin C, Patroniti N, Ranieri VM, Gattinoni L, Nava S, Terragni PP, Pesenti A, Tobin M, Mancebo J, Brochard L; PLUG Working Group (Acute Respiratory Failure Section of the European Society of Intensive Care Medicine). The application of esophageal pressure measurement in patients with respiratory failure. Am J Respir Crit Care Med. 2014 Mar 1;189(5):520-31. doi: 10.1164/rccm.201312-2193CI. PMID 24467647
- [Background] Bouhemad B, Brisson H, Le-Guen M, Arbelot C, Lu Q, Rouby JJ. Bedside ultrasound assessment of positive end-expiratory pressure-induced lung recruitment. Am J Respir Crit Care Med. 2011 Feb 1;183(3):341-7. doi: 10.1164/rccm.201003-0369OC. Epub 2010 Sep 17. PMID 20851923
- [Background] Volpicelli G, Elbarbary M, Blaivas M, Lichtenstein DA, Mathis G, Kirkpatrick AW, Melniker L, Gargani L, Noble VE, Via G, Dean A, Tsung JW, Soldati G, Copetti R, Bouhemad B, Reissig A, Agricola E, Rouby JJ, Arbelot C, Liteplo A, Sargsyan A, Silva F, Hoppmann R, Breitkreutz R, Seibel A, Neri L, Storti E, Petrovic T; International Liaison Committee on Lung Ultrasound (ILC-LUS) for International Consensus Conference on Lung Ultrasound (ICC-LUS). International evidence-based recommendations for point-of-care lung ultrasound. Intensive Care Med. 2012 Apr;38(4):577-91. doi: 10.1007/s00134-012-2513-4. Epub 2012 Mar 6. PMID 22392031
- [Background] Repesse X, Charron C, Vieillard-Baron A. Right ventricular failure in acute lung injury and acute respiratory distress syndrome. Minerva Anestesiol. 2012 Aug;78(8):941-8. Epub 2012 Jun 7. PMID 22672932
- [Background] Fichet J, Moreau L, Genee O, Legras A, Mercier E, Garot D, Dequin PF, Perrotin D. Feasibility of right ventricular longitudinal systolic function evaluation with transthoracic echocardiographic indices derived from tricuspid annular motion: a preliminary study in acute respiratory distress syndrome. Echocardiography. 2012 May;29(5):513-21. doi: 10.1111/j.1540-8175.2011.01650.x. Epub 2012 Feb 13. PMID 22324535
- [Background] Ferguson ND, Cook DJ, Guyatt GH, Mehta S, Hand L, Austin P, Zhou Q, Matte A, Walter SD, Lamontagne F, Granton JT, Arabi YM, Arroliga AC, Stewart TE, Slutsky AS, Meade MO; OSCILLATE Trial Investigators; Canadian Critical Care Trials Group. High-frequency oscillation in early acute respiratory distress syndrome. N Engl J Med. 2013 Feb 28;368(9):795-805. doi: 10.1056/NEJMoa1215554. Epub 2013 Jan 22. PMID 23339639
- [Background] Young D, Lamb SE, Shah S, MacKenzie I, Tunnicliffe W, Lall R, Rowan K, Cuthbertson BH; OSCAR Study Group. High-frequency oscillation for acute respiratory distress syndrome. N Engl J Med. 2013 Feb 28;368(9):806-13. doi: 10.1056/NEJMoa1215716. Epub 2013 Jan 22. PMID 23339638
- [Background] Terragni PP, Rosboch G, Tealdi A, Corno E, Menaldo E, Davini O, Gandini G, Herrmann P, Mascia L, Quintel M, Slutsky AS, Gattinoni L, Ranieri VM. Tidal hyperinflation during low tidal volume ventilation in acute respiratory distress syndrome. Am J Respir Crit Care Med. 2007 Jan 15;175(2):160-6. doi: 10.1164/rccm.200607-915OC. Epub 2006 Oct 12. PMID 17038660
- [Result] Ashbaugh DG, Bigelow DB, Petty TL, Levine BE. Acute respiratory distress in adults. Lancet. 1967 Aug 12;2(7511):319-23. doi: 10.1016/s0140-6736(67)90168-7. No abstract available. PMID 4143721
- [Result] ARDS Definition Task Force; Ranieri VM, Rubenfeld GD, Thompson BT, Ferguson ND, Caldwell E, Fan E, Camporota L, Slutsky AS. Acute respiratory distress syndrome: the Berlin Definition. JAMA. 2012 Jun 20;307(23):2526-33. doi: 10.1001/jama.2012.5669. PMID 22797452